CLINICAL TRIAL: NCT03194113
Title: Improving PTSD Treatments for Adults With Childhood Trauma
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Radboud University Medical Center (Other); PsyQ (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Willem Van der Does, Professor of Clinical Psychology, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P16-144
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Implosive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trauma-Focused Treatment (Active Comparator): Weekly sessions of prolonged exposure
  Interventions: Behavioral: Trauma-focused treatment
- Emotion Regulation Treatment (Active Comparator): weekly sessions of emotion regulation and skills training.
  Interventions: Behavioral: Trauma-focused treatment; Behavioral: Emotion regulation training
- Intensive Trauma-Focused Treatment (Active Comparator): prolonged exposure, 3 sessions per week
  Interventions: Behavioral: Intensive Trauma-focused treatment

INTERVENTIONS:
Behavioral: Trauma-focused treatment — Weekly sessions
  Other Names: Cognitive Behavior therapy; Prolonged exposure; Imaginal exposure
  Arms: Emotion Regulation Treatment; Trauma-Focused Treatment
Behavioral: Emotion regulation training — Managing and tolerating negative emotions, e.g. anger, sadness. Weekly sessions; preparatory to Prolonged exposure treatment
  Arms: Emotion Regulation Treatment
Behavioral: Intensive Trauma-focused treatment — Intensive version (3 sessions per week) of Trauma-focused treatment
  Other Names: Intensive Prolonged Exposure
  Arms: Intensive Trauma-Focused Treatment

SUMMARY:
The aim of this project is to investigate the effectiveness of phase-based trauma-focused therapy (PBT) and intensive trauma-focused therapy (I-TFT) for adult patients with PTSD related to childhood abuse.

We will carry out a RCT, randomizing 150 patients to receive either standard TFT, PBT or i-TFT. The effects will be assessed at two endpoints of treatment (4, 8 and 16 weeks) and after a 6 and 12 months follow-up in an intention-to-treat analysis.

DETAILED DESCRIPTION:
The Dutch treatment guidelines recommend trauma-focused treatment (TFT) for PTSD. In TFT, patients are exposed to trauma reminders that they typically avoid, until their emotional reactions decline. This treatment has been found very effective for some patients but there is much room for improvement, particularly in PTSD related to childhood abuse (CA-PTSD). Symptom exacerbation, non-attendance and dropout rates of up to 40% have been observed in patients with CA-PTSD.

Two alternative treatments have been proposed. Firstly, TFT may be preceded by emotion regulation and interpersonal skills training. This is called phase-based treatment (PBT). The rationale is that patients with CA-PTSD have affect regulation and interpersonal problems that interfere with effective delivery of TFT. These problems are rooted in the detrimental developmental effects of abuse (often by an attachment figure). PBT indeed resulted in more favorable outcomes and fewer dropouts. In international guidelines, PBT was recently recommended as treatment of choice for patients with CA-PTSD and comorbidity.

Another innovative treatment is intensive TFT (i-TFT), which means delivering TFT in 4 instead of 16 weeks. The condensed format enhances learning and prevents the buildup of anticipatory anxiety, which in turn affects the patients' motivation. Patients with CA-PTSD are also characterized by high psychosocial stressors, leading to problems with treatment attendance and compliance. The condensed format may improve motivation, attendance and compliance. I-TFT was recently tested in a case series in patients with CA-PTSD and in a randomized controlled trial (RCT) with patients with adulthood-related PTSD. Both studies had very low dropout rates (0-3%) and fast recovery.

The aim of the current study is to investigate the (cost)effectiveness of two innovative forms of trauma-focused therapy for patients with CA-PTSD: phase-based therapy (emotion regulation skills training followed bij PE) and intensive PE (i-PE). The effects will be assessed post-treatment and after a 6 and 12 months follow-up in an intention-to-treat analysis. Results will be disseminated and included in treatment guidelines. The ultimate goal is to improve quality of care and contribute to treatment innovation for this severely ill target population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD according to DSM-5, including at least one specific discrete memory of a traumatic event
* Multiple traumata related to childhood sexual/physical abuse that occurred before 18 years of age, and committed by a primary caretaker or an authority figure as index event
* Symptom severity: CAPS score > 25
* Sufficient fluency in Dutch to complete the treatment and research protocols

Exclusion Criteria:

* Involved in legal procedures concerning admission or stay in The Netherlands
* Involvement in compensation issues
* Pregnancy
* Severe non-suicidal self-injury (NSSI) in the last two months (hospital referral required)
* Suicidality in the last 2 months
* Alcohol or drug dependence in last 2 months
* Cognitive impairment (estimated IQ < 70)
* Changes in psychotropic medication in the two months prior to inclusion
* Current psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity | 16 weeks
  Clinician Administered Posttraumatic Stress Inventory (CAPS-5) total score

SECONDARY OUTCOMES:
Depressive symptom severity | 16 weeks
  total score on Inventory of Depressive Symptomatology (IDS)
Quality of Life score | 16 weeks
  EQ5D5L total score
Responder rate | 16 weeks
  Meeting pre-defined criteria for remission
Dropout rate | 16 weeks
  premature termination of treatment by patient
Emotion regulation | 16 weeks
  ICD-11 Trauma Questionnaire and Difficulties in Emotion Regulation Scale (DERS)
Self-reported PTSD symptoms | 16 weeks
  Post-traumatic Stress Disorder Checklist (PCL-5)
Interpersonal difficulties | 16 weeks
  ICD-11 Trauma Questionnaire and Inventory of Interpersonal Problems (IIP)
Self-concept | 16 weeks
  ICD-11 Trauma Questionnaire and Rosenberg self-esteem scale (RSS)

CONTACTS AND LOCATIONS:
Overall Officials: Willem Van Der Does, PdhD, Study Chair — head of department of clinical psychology
Locations (2):
- Netherlands (2):
  - Leiden University - Institute of Psychology, Leiden, South Holland
  - PsyQ department of psychotrauma, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported from this study may be shared, after deidentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Zayfert C, Deviva JC, Becker CB, Pike JL, Gillock KL, Hayes SA. Exposure utilization and completion of cognitive behavioral therapy for PTSD in a "real world" clinical practice. J Trauma Stress. 2005 Dec;18(6):637-45. doi: 10.1002/jts.20072. PMID 16382429
- [Background] Hendriks, L., & Van Minnen, A. (2014). What to do with treatment failures: Intensive (Prolonged) Exposure treatment for PTSD. Presentation at EABCT Conference The Hague.
- [Background] Ehlers A, Hackmann A, Grey N, Wild J, Liness S, Albert I, Deale A, Stott R, Clark DM. A randomized controlled trial of 7-day intensive and standard weekly cognitive therapy for PTSD and emotion-focused supportive therapy. Am J Psychiatry. 2014 Mar;171(3):294-304. doi: 10.1176/appi.ajp.2013.13040552. PMID 24480899
- [Background] Cloitre M, Stovall-McClough KC, Nooner K, Zorbas P, Cherry S, Jackson CL, Gan W, Petkova E. Treatment for PTSD related to childhood abuse: a randomized controlled trial. Am J Psychiatry. 2010 Aug;167(8):915-24. doi: 10.1176/appi.ajp.2010.09081247. Epub 2010 Jul 1. PMID 20595411
- [Background] Cloitre, M., Courtois, C.A., Ford, J.D., Green, B.L., Alexander, P., Briere, J. et al. (2012). The ISTSS Expert Consensus Treatment Guidelines for Complex PTSD in Adults. http://www.istss.org/AM/Template.cmf?Section=ISTSS_Complex_PTSD_Treatment_Guidelines&Template=/CM/ContentDisplay.cfm&ContentID=5185
- [Derived] Oprel DAC, Hoeboer CM, Schoorl M, de Kleine RA, Cloitre M, Wigard IG, van Minnen A, van der Does W. Effect of Prolonged Exposure, intensified Prolonged Exposure and STAIR+Prolonged Exposure in patients with PTSD related to childhood abuse: a randomized controlled trial. Eur J Psychotraumatol. 2021 Jan 15;12(1):1851511. doi: 10.1080/20008198.2020.1851511. eCollection 2021. PMID 34630934
- [Derived] Oprel DAC, Hoeboer CM, Schoorl M, De Kleine RA, Wigard IG, Cloitre M, Van Minnen A, Van der Does W. Improving treatment for patients with childhood abuse related posttraumatic stress disorder (IMPACT study): protocol for a multicenter randomized trial comparing prolonged exposure with intensified prolonged exposure and phase-based treatment. BMC Psychiatry. 2018 Dec 12;18(1):385. doi: 10.1186/s12888-018-1967-5. PMID 30541492